CLINICAL TRIAL: NCT00537251
Title: 32-Week, Open, Randomized, Cross-Over, Local, Multicenter Clinical Trial Comparing Insulin Glargine in Combination With Insulin Analogue (Insulin Lispro) to NPH Insulin in Combination With Regular Insulin in Type 1 Diabetes Mellitus Patients in an Intensified Insulin Regimen.
Brief Title: 32 Week, Open, Randomized, 2 Way Cross Over Multicentre Trial to Compare Safety & Efficacy of Combination of HOE901 Insulin Analogue Once Daily at Bedtime + Lispro Insulin Before Meals vs NPH Insulin (Twice a Day) + Regular in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4023
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2007-10-01 (Estimated); Status verified 2007-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin glargine

SUMMARY:
To compare the efficacy (in terms of metabolic control evaluated through HbA1c levels) of treatment with insulin glargine as basal insulin and insulin analogue (insulin lispro) as mealtime insulin with a regimen of insulin NPH as basal insulin with regular insulin, as mealtime insulin, after a 16 week treatment phase with each regimen and to compare the safety of both treatments, evaluated through hypoglycemic rates.

DETAILED DESCRIPTION:
Multicenter, open-label, randomized (allocation ratio 1:1), cross-over with two treatment phases of 16 weeks each in two treatment groups:

* Study arm with insulin glargine + insulin lispro (phase 1) and insulin NPH + regular insulin (phase 2)
* Insulin NPH + regular insulin (phase 1) and insulin glargine + insulin lispro (phase 2)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 1 diabetes mellitus
* 18-65 years of age
* C-Peptide negative
* Treated at least for 6 months with multiple daily doses of insulin and with HbA1c greater than or equal to 7.0% and less than or equal to 9.5% and a BMI less than or equal to 35 kg/m².
* Women of childbearing potential must have a negative pregnancy test in visit 1 and must use an effective contraceptive method during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-11; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Compare efficacy of insulin glargine & short acting insulin (Lispro), NPH insulin regime as basal insulin and regular insulin for meal insulin for metabolic control, evaluated by means of HbA1c . | after 16 weeks of treatment with each treatment regime

CONTACTS AND LOCATIONS:
Overall Officials: Jose Taboada Mosquera, Study Director — Sanofi